CLINICAL TRIAL: NCT00822445
Title: Diagnostic Value and Prognostic Value of the Blood Level Determination of S100 Protein in Minor or Mild Traumatic Brain Injury (GCS Glasgow Score 9 to 15).
Brief Title: S100 Protein in Minor/Mild Traumatic Brain Injury
Acronym: S100
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: IC0601
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2008-02

CONDITIONS: Minor/Mild Traumatic Brain Injury
Keywords: Biomarker; S100 protein; Traumatic brain injury; Craniocerebral tomodensitometry; Neurological sequelae
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Traumatic brain injury (TBI) is a Public Health problem, because of the numbers of events (more than 200,000 per year in France). Craniocerebral tomodensitometry (CCT) is widely used for the diagnosis of minor/mild TBI, but both the access to the CCT and the cost of this imagery are critical factors. We hypothesized that the blood level measurement of S100 protein (S100), a neurological biomarker of cerebral injury, would help to the clinical evaluation of minor/mild head injury events, and would be an economic alternative to CCT for the diagnosis of these pathologies. In addition, a part of the study will explore the prognostic value of such blood level S100 determination for the evaluation of medical/social consequences of minor/mild TBI.

Medical objective of the study:

1. to assess the contribution of early determination (to medical care) of S100 for the diagnosis of minor/moderate TBI (TCCMM - Glasgow sup or equal to 9),
2. to determine the usefulness of a second dosage three hours later for the medical decision.

In other words, to compare S100 biomarker and CCT considered as a reference ( "Gold Standard") for the diagnosis or exclusion of TCCMM, and to precise its terms of use.

Economic objective:

to conduct a cost-effectiveness study of blood level determination of S100 vs. CCT for the diagnosis of minor/moderate TBI and its medical/social consequences

DETAILED DESCRIPTION:
Nearly two hundred thousand head injury cases (Traumatic Brain Injury - TBI) are reported each year in France. Less than 5% are severe, defined by a Glasgow score (GCS) above 9. Epidemiological studies indicate that TBI is the fourth leading cause of death and disability in industrialized countries. Major causes of mild/minor TBI are falls and domestic trauma in the elderly or children, and sports accidents. The minor/mild brai injury (MBI) may represent 5 to 10% of emergency consultations in the UAA.

The severity of a head injury is assessed by the Glasgow Coma Scale (GCS), and TBI are divided into three groups: minor (13-15), moderate (9-12) , severe (3-8). Definition of TCC has considerably evolved over the past 20 years, to take into account the pathophysiologic lesions secondary is related to systemic factors (hypotension, hypoxia ...) and intracranial factors ( intracranial hypertension, seizures committals ...). These side events, occurring within hours or days after the primary injury caused by an impact (contusion, hematoma, deceleration), increase the morbidity of the initial event, and must therefore be detected both early and fully.

The diagnosis of TBI requires imaging data such as craniocerebral tomography (CCT), which will be renewed after 24 hours and if necessary the following day. Until now, no pertinent biological marker was proposed to complete the clinical/imagery investigation of mild/moderate TBI.

S100B protein (S100) is a constitutive protein of glial cells, whose physiological functions are both intracellular, i.e. intracytosolic calcium binding, and extracellular, e.g. by promoting neuritic proliferation and/or neuronal apoptosis. Due to specificity of its cellular expression, S100B protein is a useful biological marker of acute neurological disorders, such as ischemic or haemorrhagic stroke, and traumatic head injury. hemorrhage, ischemic stroke) or traumatic (TCC). Plasma S100 is significantly increased in subjects with a major TCC, but also in the majority of minor or moderate TBI. A prognostic value of S100 also was suggested : patients who exhibited medical or social sequelae after several months after TBI also shoed high plasma levels of S100 in the first hours of the head injury. Such results of international clinical studies proposed S100 as a biomarker of diffuse brain injury, and indicate the importance of early determination of plasma concentration of S100 and its integration among the other elements of diagnosis (imaging) for assessing the severity of trauma and its short and long terms.

Medical objective of the study:

1. to assess the contribution of early determination (to medical care) of S100 for the diagnosis of minor/moderate TBI (TCCMM - Glasgow sup or equal to 9),
2. to determine the usefulness of a second dosage three hours later for the medical decision.

In other words, to compare S100 biomarker and CCT considered as a reference ( "Gold Standard") for the diagnosis or exclusion of TCCMM, and to precise its terms of use.

Economic objective:

to conduct a cost-effectiveness study of blood level determination of S100 vs. CCT for the diagnosis of minor/moderate TBI and its medical/social consequences.

ELIGIBILITY:
Inclusion criteria :

* Patient with suspected minor/mild TBI justifying a cerebral tomodensitometry (blow to the head, concussion ± treatment by AVK or antiaggregants
* Age above 65 years ± temporary loss of consciousness [<10 minutes] ±amnesia ± major headache ±vomiting
* Glasgow score at admission sup or equal to 9
* Admission within 3 hours after to the traumatic event
* Cerebral tomodensitometry within 6 hours after admission
* Informed consent of the subject

Exclusion criteria :

* Age <18 or> 80 years
* Glasgow score at admission <9
* No prescription of cerebral tomodensitometry
* Multiple, fractures
* Pregnancy
* Acute (meningitis...) or chronic (encephalitis, all neurodegenerative diseases ...) neurological disease
* Renal failure (creatinine> 130 µmol/L)
* Malignant melanoma
* Loss of consciousness> 10 minutes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Minor/mild traumatic brain injury
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2008-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Relationship between S100 levels and the diagnosis of minor/moderate TBI by craniocerebral tomodensitometry | during the study

SECONDARY OUTCOMES:
Positive and negative predictive values of S100 level for the diagnosis and the prognosis of minor/moderate TBI | during the study

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Beaudeux, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Groupe Hospitalier Pitié-Salpêtrière - Charles Foix, Ivry-sur-Seine, France